CLINICAL TRIAL: NCT06234241
Title: Normal Reference Values of Cardiac Measurements by Echocardiography in Chinese Han Adults Based on Artificial Intelligence: A Multi-center Study in China
Brief Title: Normal Values of Cardiac Measurements by Echocardiography in Chinese Based on Artificial Intelligence
Status: Completed | Type: Observational
Sponsor: Tianxin Dong (Other)
Responsible Party: Sponsor-Investigator, Tianxin Dong, MD, First Hospital of China Medical University
Organization: First Hospital of China Medical University (Other)
Other Study IDs: 2023-445
Record Dates: First submitted 2024-01-23; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Heart Chambers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Echocardiography — Echocardiography was performed in all enrolled populations.

SUMMARY:
Establish echocardiographic normal reference values of Chinese Han adults based on artificial intelligence.

DETAILED DESCRIPTION:
We will establish normal reference values for the volume, function and strain of various heart chambers of Chinese people based on the recruitment of healthy Chinese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years; No history or clinical evidence of cardiac, cardiovascular, lung, or kidney disease; No abnormal findings on physical examination, biochemical examination, electrocardiography, or echocardiography.

Exclusion Criteria:

* Hypertension (blood pressure [BP] > 140/80 mmHg) or receiving medication for hypertension; body mass index > 30 kg/m2; total cholesterol ≥ 6.2 mmol/L, triglyceride ≥ 2.3 mmol/L, or high-density lipoprotein cholesterol < 1.0 mmol/L; endocrine diseases, such as diabetes mellitus (fasting blood glucose ≥ 7.0 mmol/L), thyroid disease, pheochromocytoma, adrenal insufficiency, and hyperaldosteronism; anemia; abnormal liver function; connective tissue diseases, such as rheumatoid arthritis, vasculitis, systemic lupus erythematosus, dermatomyositis, and scleroderma; malignancy; current pregnancy or lactation; professional sport activity; and a history of alcoholism.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Chinese Han healthy adults
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Cardiac volumes | 2024-10-31
  Including the left and right atria and left and right ventricles
Cardiac Function | 2024-10-31
  Including the left and right atria and left and right ventricles
Cardiac strain | 2024-10-31
  Including the left and right atria and left and right ventricles

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided